CLINICAL TRIAL: NCT06456606
Title: The Effect of Prone Position on Right Ventricular Functions in CARDS: is Survival Predictable When Evaluated Through Transesophageal Echocardiography?
Brief Title: Cardiopulmonary Effects of Prone Position in CARDS
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Dicle Birtane, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2022/40
Record Dates: First submitted 2024-05-31; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: ARDS Due to Disease Caused by SARS Co-V-2; Right Ventricular Dysfunction
Keywords: transesophageal echocardiography; cards; heart lung interactions; prone position; right ventricle
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group a: 30 moderate-to-severe C-ARDS patients who were treated with prone position in the first 48 hours of invasive mechanical ventilation support. It was evaluated with transesophageal echocardiography three times: before prone position (T0), the first hour of prone position (T1), and the first hour of returning to the supine position (T0 + 24 hours) (T2) after 23 hours prone position treatment.
  Interventions: Procedure: before prone position; Procedure: the first hour of prone position; Procedure: the first hour of returning to the supine position

INTERVENTIONS:
Procedure: before prone position — It was evaluated with transesophageal echocardiography
  Other Names: t0
Procedure: the first hour of prone position — It was evaluated with transesophageal echocardiography
  Other Names: t1
Procedure: the first hour of returning to the supine position — It was evaluated with transesophageal echocardiography
  Other Names: t2

SUMMARY:
In coronavirus disease-2019 (COVID-19)-related ARDS (C-ARDS), especially in the severe form, increased shunt rate, impaired ventilation/perfusion ratio (V/Q), hypoxic pulmonary vasoconstriction inhibition, and increased immune microthrombosis may have similar effects on the right ventricle .The cardiopulmonary pathophysiology and outcomes of C-ARDS vary, and this variability requires monitoring to follow the diagnosis and treatment process. This study aimed to increase the treatment success of the prone position in C-ARDS and to provide a prognostic factor for survival by analyzing and monitoring heart-lung interactions. Therefore, we used transesophageal echocardiography (TEE) to evaluate the cardiopulmonary effects of prone position.

DETAILED DESCRIPTION:
This prospective study included 30 moderate-to-severe C-ARDS patients who were treated with prone position in the first 48 hours of invasive mechanical ventilation support. It was evaluated with transesophageal echocardiography three times: before prone position (PP) (T0), the first hour of PP (T1), and the first hour of returning to the supine position (T0 + 24 hours) (T2) after 23 hours prone position treatment. Right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA) was preferred right ventricular evaluations as primer outcome. Static compliance (C-stat) was examined in the evaluation of the pulmonary effect of prone position as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Patients diagnosed with polymerase chain reaction/computed tomography results
* Moderate/severe severity class according to the Berlin ARDS classification
* Prone position applied in the first 48 h after orotracheal intubation in treatment
* Obtaining an informed consent form

Exclusion Criteria:

* Pulmonary embolism
* Pneumothorax
* Heart valve disease
* Pregnancy
* Perforated esophageal varices
* Coagulopathy
* Esophageal stricture
* Esophageal tumor
* Neck fracture
* Thrombocytopenia
* Gastrointestinal bleeding
* Previous stomach surgery
* Previous esophageal surgery
* Esophageal perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate/severe C-ARDS patients admitted to the Bakırköy Dr Sadi Konuk Training and Research Hospital Anesthesiology and Reanimation Clinic Intensive Care Unit, who received invasive mechanical ventilation support and applied prone position in the first 48 h were included.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA) change during prone position. | It was evaluated with transesophageal echocardiography three times: before prone position (T0), the first hour of prone position (T1), and the first hour of returning to the supine position (T0 + 24 hours) (T2) after 23 hours prone position treatment
  It was preferred right ventricular recovery evaluation.

SECONDARY OUTCOMES:
Static compliance (C-stat) change with prone position | It was evaluated with transesophageal echocardiography three times: before prone position (T0), the first hour of prone position (T1), and the first hour of returning to the supine position (T0 + 24 hours) (T2) after 23 hours prone position treatment
  It was examined in the evaluation of the pulmonary effect of prone position as secondary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data available from the publication date can start If requested, data will be shared with medical doctors dealing with
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Fossali T, Pavlovsky B, Ottolina D, Colombo R, Basile MC, Castelli A, Rech R, Borghi B, Ianniello A, Flor N, Spinelli E, Catena E, Mauri T. Effects of Prone Position on Lung Recruitment and Ventilation-Perfusion Matching in Patients With COVID-19 Acute Respiratory Distress Syndrome: A Combined CT Scan/Electrical Impedance Tomography Study. Crit Care Med. 2022 May 1;50(5):723-732. doi: 10.1097/CCM.0000000000005450. Epub 2022 Apr 11. PMID 35200194
- [Result] Evrard B, Goudelin M, Fedou AL, Vignon P. Hemodynamic response to prone ventilation in COVID-19 patients assessed with 3D transesophageal echocardiography. Intensive Care Med. 2020 Nov;46(11):2099-2101. doi: 10.1007/s00134-020-06217-w. Epub 2020 Aug 26. No abstract available. PMID 32844261
- [Result] Beyls C, Daumin C, Hermida A, Booz T, Ghesquieres T, Crombet M, Martin N, Huette P, Jounieaux V, Dupont H, Abou-Arab O, Mahjoub Y. Association between the Right Ventricular Longitudinal Shortening Fraction and Mortality in Acute Respiratory Distress Syndrome Related to COVID-19 Infection: A Prospective Study. J Clin Med. 2022 May 6;11(9):2625. doi: 10.3390/jcm11092625. PMID 35566751
- [Result] Temperikidis P, Koroneos A, Xourgia E, Kotanidou A, Siempos II. Abnormal Right Ventricular Free Wall Strain Prior to Prone Ventilation May Be Associated With Worse Outcome of Patients With COVID-19-Associated Acute Respiratory Distress Syndrome. Crit Care Explor. 2022 Jan 11;4(1):e0620. doi: 10.1097/CCE.0000000000000620. eCollection 2022 Jan. PMID 35036925
- [Result] Tonetti T, Grasselli G, Rucci P, Alessandri F, Dell'Olio A, Boscolo A, Pasin L, Sella N, Mega C, Melotti RM, Girardis M, Busani S, Bellani G, Foti G, Grieco DL, Scaravilli V, Protti A, Langer T, Mascia L, Pugliese F, Cecconi M, Fumagalli R, Nava S, Antonelli M, Slutsky AS, Navalesi P, Pesenti A, Ranieri VM. Synergistic Effect of Static Compliance and D-dimers to Predict Outcome of Patients with COVID-19-ARDS: A Prospective Multicenter Study. Biomedicines. 2021 Sep 15;9(9):1228. doi: 10.3390/biomedicines9091228. PMID 34572414